CLINICAL TRIAL: NCT06736275
Title: A Phase I Study on Evaluating the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of SXRN Plasmid DNA Technique in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jiangsu Nutai Biologics Co., Ltd (Industry)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AA0101
Record Dates: First submitted 2024-12-01; First posted 2024-12-16 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-08

CONDITIONS: Advanced Cancer; Cachexia
Keywords: micoRNA
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Intervention Model Description: Accelerated titration and "3+3" dose escalation: This study plans to start dose escalating from 2 mg, followed by 4 mg, and 10 mg as tentatively designated escalating dose groups. An "accelerated titration" strategy will be implemented in the early dose escalation phase (2 mg dose group) in this study, with only 1 subject enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group (Experimental): In this study, three dose levels are initially formulated, namely 2mg, 4mg, and 10mg of SXRN, adopting an accelerated titration followed by the traditional "3+3" design. The first day of infusion for each dose is referred to as C1D1, with the administration of QD for 5 consecutive days, followed by a 2-day break; Each treatment cycle will last 3 weeks (21 days), and the subsequent infusion regimen, including interval, frequency and dose, may be adjusted based on the initial safety and PK parameters.
  Interventions: Drug: SXRN

INTERVENTIONS:
Drug: SXRN — SXRN is a naked plasmid DNA drug targeting miRNA. Accelerated titration and "3+3" dose escalation:In light of ethical considerations and with the aim of minimizing the number of patients possibly exposed to potentially ineffective doses, an "accelerated titration" strategy will be implemented in the early dose escalation phase (2 mg dose group) in this study, with only 1 subject enrolled. If no DLT occurs to the 3 subjects under the given dose in the DLT valuation window (the 1st cycle, 3 weeks), the study will proceed to the next dose (dose escalation in the same subject is not allowed); if one subject develops DLT, 3 additional subject s will be included to the current dose group; if ≥2 DLTs occur in the dose group with 3 or 6 subject s, the dose escalation will be stopped. The decision is made by discussion among the investigators whether to terminate the escalation or consider adjusting the dose for exploration.

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and tolerability of SXRN Plasmid DNA Technique in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase I, open-label, dose-escalation study to investigate the safety, tolerability, pharmacokinetics and preliminary efficacy of SXRN Plasmid DNA Technique in patients with advanced solid tumors. Three dose levels are initially formulated, namely 2mg, 4mg, and 10mg of SXRN, adopting an accelerated titration followed by the traditional "3+3" design. SXRN will be administered daily x 5 with 2 days off (total of 21 days) for 3 weeks followed by a no-treatment observation period.

ELIGIBILITY:
Inclusion Criteria:

* male or female, aged 18~75 at the time of signing the ICF;
* patient with advanced solid tumors who have failed/cannot tolerate previous standard therapies or lack conventional effective therapies;
* at least one measurable or evaluable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1);
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
* expected survival time ≥12 weeks;
* lab results and organ function tested within 7 days before the initial infusion meet the criteria below:
* Blood routine: 1)Absolute Neutrophil Count (ANC) ≥1.5×10^9/L;2)Platlets (PLT) Count≥90×10^9/L; 3)Hemoglobins (Hb) ≥90 g/L.

Note: the criteria above shall still be maintained within 14 days before the initial infusion, either without the need of blood transfusion, or using supportive treatment including granulocyte colony-stimulating factor (G-CSF), thrombopoietin (TPO), interleukin-11 (IL-11), and erythropoietin (EPO), and etc.

* Blood biochemistry: 1)Total bilirubin (TBIL) ≤3.0 × upper limit of normal (ULN); 2)Serum creatinine (SCr) ≤1.5 × ULN or creatinine clearance (CrCl) by Cockroft Gault formula ≥50 mL/min; 3)Aspartate Amino Transferase (AST), Alanine Aminotransferase (ALT) ≤2.5×ULN; for participants with liver metastasis, AST, ALT≤5.0×ULN, and ALP≤6.0×ULN; d)Albumin (ALB) ≥30g/L.
* Urine protein ≤2+ (if >2+, urine protein shall be collected for 24 hours; total protein ≤1g is acceptable for inclusion).
* International Normalized Ratio (INR), Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN.

Note: for subjects receiving precautious anti-coagulation treatment, the investigator shall determine whether INR and APTT remains in a safe and effective range for treatment.

* Left Ventricular Ejection Fraction (LVEF) ≥50%.
* can understand and voluntarily sign the Informed Consent Form (ICF); must be voluntary and able to finish the study program and follow-up tests.

Exclusion Criteria:

* Subjects who meet any of the criteria below must not be included:
* has received any of the anti-tumor treatments below:a) received cytotoxic chemotherapy, tumor immunotherapy, anti-tumor biologics or other trail agents within 4 weeks or 5 half-times (whichever is shorter) before the initial infusion.b)received an oral small-molecule targeted anti-tumor agent within 2 weeks before the first infusion or for five half-lives(whichever was shorter).c) received anti-tumor Chinese patent medicine approved by NMPA within 2 weeks before the initial infusion.d) received more than 30% bone marrow radiotherapy or large area radiotherapy within 2 weeks before initial infusion (palliative radiotherapy at the bone or superficial lesions is acceptable).
* participated in and received an investigational drug or device clinical trial within 4 weeks before initial infusion.
* Patients who had undergone or planned to undergo major surgery or interventional therapy (excluding tumor biopsy, puncture, etc.) within 4 weeks before initial infusion.
* unrecovered from the toxic reaction caused by previous anti-tumor treatment (not recovered to ≤ grade 1 or baseline; not including toxic reactions with no safety risk as determined by the investigator, such as alopecia, asymptomatic hypothyroidism caused by immune checkpoint inhibitors that can be treated with only thyroid hormone and remains stable, and etc.).
* with clinically uncontrollable serous effusion (pleural effusion, ascites and pericardio effusion). Conditions may include: moderate or above sized effusion, received within 2 weeks before the selection or plans to receive local treatments (including drainage, peritoneal shunt, and cell-free concentrated ascites reinfusion, and etc.), or effusion obviously increased within 2 weeks after the local treatment and thus needs long-term catherterization. Candidates who meet any of the conditions above, or determined by the investigator as unsuitable, shall not be included.
* with central nervous system metastasis and show relating symptoms.
* with a history of other malignant tumors, except for those that have received radical surgery and not relapsed 5 years thereafter, such as carcinoma in situ of cervix, skin basal cell carcinoma, and etc.
* with a history of immune deficiency diseases, including acquired or congenital immunodeficiency disorders; or a history of organ transplantation, heterogeneous bone marrow transplantation, or autologous hematopoietic stem cell transplantation.
* had (non-infectious) lung inflammation / interstitial lung disease that required steroid treatment within 4 weeks before the initial infusion.
* with a history of severe cardiovascular and cerebrovascular diseases, including but not limited to:

  1. severe abnormalty in cardiac rhythm or conduction, such as ventricular arrhythmia requiring clinical intervention, atrioventricular block of II~III grade, and etc.;
  2. cardiac insufficiency of III~IV grade as defined by New York Heart Association(NYHA);
  3. acute coronary syndrome, congestive cardiac failure, aortic dissection, cerebral stroke or other grade 3 or above cardio-cerebral vascular events within 6 months before the initial infusion.
* with uncontrollable high blood pressure (systolic pressure ≥160 mmHg and/or diastolic pressure ≥100 mmHg) after treatment with anti-hypertensive drugs of stable doses.
* with active chronic hepatitis B (such as, HbsAg or HbcAb positive and HBV DNA ≥ lower limit of detection, active hepatisis C (such as, HCV antibody positive and HCV RNA≥ lower limit of detection), or HIV infection.
* with active infections within 2 weeks before the initial infusion that require systematic treatment.
* with a history of active tuberculosis infection within 1 year before the initial infusion.
* had or has uncontrollable or serious diseases that may interfere with the participation or evaluation in the study, as considered by the investigator;
* known to be allergic or taking drugs contradictionary to the study drug (Suplussirna) or its excipients.
* premenopause female candidates (postmenopausal female patients can only be considered infertilewhen they have been postmenopausal for at least 12 months) with positive results in serum pregnancy test; candidates of reproductive age (also including female spouse of reproductive age of male candidates), during the study or within 6 months after the last infusion, who will probably bear children, breastfeed, or are unwilling to cake effective contraceptives, as considered by the investigator.
* other conditions that are determined by the investigator as unsitable for entering this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Recommended Dose for Expansion (RDE) of SXRN | 12 months
  To determine the Maximum Tolerated Dose (MTD) and Recommended Dose for Expansion (RDE) of SXRN in the treatment of advanced solid tumors

SECONDARY OUTCOMES:
Pharmacokinetic parameters of SXRN | 12 months
  Maximum plasmid Concentration [Cmax]
Preliminary anti-tumor efficacy of SXRN | 12 months
  Anti-tumor activity: objective remission rate (ORR), duration of remission (DOR), disease control rate (DCR), time to remission (TTR) and progression free survival (PFS) basing on RECIST v1.1; overall survival (OS);
Weight improvement of SXRN in patients with advanced solid tumors | 12 months
  Body weight
Appetite improvement of SXRN in patients with advanced solid tumors | 12 months
  Change in patient's quality of life on the FAACT-A/ CS-12 questionnaire (score)
Pain alleviating efficacy of SXRN in patients with advanced solid tumors | 12 months
  Change in patient's quality of life on the numeric rate scale (NRS) questionnaire (score)

OTHER OUTCOMES:
the SXRN transcripts,its targets, and possible regulated targets | 12 months
  Explore the expression changes of the following indicators:the SXRN transcripts 1-RNA, Its targets -miR-214, possible regulated targets-A2AR, INSL3, and Inflammatory Biomarkers

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Garcia GE, Truong LD, Chen JF, Johnson RJ, Feng L. Adenosine A(2A) receptor activation prevents progressive kidney fibrosis in a model of immune-associated chronic inflammation. Kidney Int. 2011 Aug;80(4):378-88. doi: 10.1038/ki.2011.101. Epub 2011 Apr 20. PMID 21508927
- [Background] Wang Q, Liu Y, Wu Y, Wen J, Man C. Immune function of miR-214 and its application prospects as molecular marker. PeerJ. 2021 Feb 16;9:e10924. doi: 10.7717/peerj.10924. eCollection 2021. PMID 33628646
- [Background] Zhao L, Liu YW, Yang T, Gan L, Yang N, Dai SS, He F. The mutual regulation between miR-214 and A2AR signaling plays an important role in inflammatory response. Cell Signal. 2015 Oct;27(10):2026-34. doi: 10.1016/j.cellsig.2015.07.007. Epub 2015 Jul 11. PMID 26171727
- [Background] Takayama K, Atagi S, Imamura F, Tanaka H, Minato K, Harada T, Katakami N, Yokoyama T, Yoshimori K, Takiguchi Y, Hataji O, Takeda Y, Aoe K, Kim YH, Yokota S, Tabeta H, Tomii K, Ohashi Y, Eguchi K, Watanabe K. Quality of life and survival survey of cancer cachexia in advanced non-small cell lung cancer patients-Japan nutrition and QOL survey in patients with advanced non-small cell lung cancer study. Support Care Cancer. 2016 Aug;24(8):3473-80. doi: 10.1007/s00520-016-3156-8. Epub 2016 Mar 22. PMID 27003901
- [Background] Fearon KC, Voss AC, Hustead DS; Cancer Cachexia Study Group. Definition of cancer cachexia: effect of weight loss, reduced food intake, and systemic inflammation on functional status and prognosis. Am J Clin Nutr. 2006 Jun;83(6):1345-50. doi: 10.1093/ajcn/83.6.1345. PMID 16762946
- [Background] Malik M, Michalak M, Radecka B, Gelej M, Jackowska A, Filipczyk-Cisarz E, Hetman K, Foszczynska-Kloda M, Kania-Zembaczynska B, Manka D, Orlikowska M, Rogowska-Dros H, Bodnar L. Prognostic Value of Sarcopenia in Metastatic Colorectal Cancer Patients Treated with Trifluridine/Tipiracil. J Clin Med. 2021 Oct 30;10(21):5107. doi: 10.3390/jcm10215107. PMID 34768626
- [Background] Argiles JM, Busquets S, Stemmler B, Lopez-Soriano FJ. Cancer cachexia: understanding the molecular basis. Nat Rev Cancer. 2014 Nov;14(11):754-62. doi: 10.1038/nrc3829. Epub 2014 Oct 9. PMID 25291291
- [Background] Loberg RD, Bradley DA, Tomlins SA, Chinnaiyan AM, Pienta KJ. The lethal phenotype of cancer: the molecular basis of death due to malignancy. CA Cancer J Clin. 2007 Jul-Aug;57(4):225-41. doi: 10.3322/canjclin.57.4.225. PMID 17626119
- [Background] Scarpi E, Maltoni M, Miceli R, Mariani L, Caraceni A, Amadori D, Nanni O. Survival prediction for terminally ill cancer patients: revision of the palliative prognostic score with incorporation of delirium. Oncologist. 2011;16(12):1793-9. doi: 10.1634/theoncologist.2011-0130. Epub 2011 Oct 31. PMID 22042788
- [Background] Mondello P, Mian M, Aloisi C, Fama F, Mondello S, Pitini V. Cancer cachexia syndrome: pathogenesis, diagnosis, and new therapeutic options. Nutr Cancer. 2015;67(1):12-26. doi: 10.1080/01635581.2015.976318. Epub 2014 Dec 16. PMID 25513730